CLINICAL TRIAL: NCT06535685
Title: A Single-centre, Prospective, Open-label, Single-arm Study of Romiplostim for the Treatment of Refractory Transfusion-dependent Non-severe Aplastic Anaemia (NSAA)
Brief Title: A Study of Romiplostim for the Treatment of Refractory Transfusion-dependent NSAA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, chief physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRA-2024-002
Record Dates: First submitted 2024-07-24; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — romiplostim

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Romiplostim group (Experimental): Romiplostim group
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Enrolled patients will be given Romiplostim (20 µg/kg subcutaneously once a week) for a minimum of 3 months.

SUMMARY:
Efficacy and safety of Romiplostim in the treatment of refractory transfusion-dependent NSAA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Diagnosis consistent with refractory transfusion dependence NSAA defines refractory as patients who have failed to respond to at least 6 months of prior first-line treatment with adequate doses of cyclosporine (3-5 mg/kg) and who have been treated with an adequate dose of at least one povidone for 3 months. Definition of transfusion dependence: at least 1 component transfusion on average every 8 weeks and duration of transfusion dependence ≥ 4 months.
3. Satisfy at least one of the following conditions at the time of enrolment: haemoglobin <90 g/L, platelets <30×10^9/L, neutrophils <1.0×10^9/L.
4. Agree to sign the consent form.
5. An Eastern Cooperative Oncology Group (ECOG) score of 0-2.

Exclusion Criteria:

1. Other causes of whole blood cytopenia, such as myelodysplastic syndromes (MDS).
2. Presence of cytogenetic evidence of clonal haematological bone marrow disorders (MDS, AML).
3. PNH clones ≥50%.
4. Haematopoietic stem cell transplantation (HSCT) prior to enrolment.
5. Prior treatment with ATG.
6. Infection or haemorrhage uncontrolled by standard therapy.
7. Allergy to roprostin.
8. Active HIV, HCV or HBV infection or cirrhosis or portal hypertension.
9. Any concomitant malignancy, localised basal cell carcinoma of the skin within 5 years.
10. Liver and renal function at baseline that is more than two times normal.
11. Active infection.
12. Past history of thromboembolic events, heart attack or stroke (including antiphospholipid antibody syndrome) and current use of anticoagulants.
13. Pregnant or lactating (breastfeeding) women.
14. Participation in another clinical trial within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-02 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 months
  Overall response rate (ORR) was defined as the ratio of complete response (CR) + partial response (PR).CR was defined as a haemoglobin level ≥120 g/L, neutrophil count >1.5 × 10^9/L and platelet count >150 × 10^9/L in patients who did not receive a transfusion.PR was defined as not being transfusion-dependent (if previously transfusion-dependent), or doubling or normalisation of at least one cell line or baseline increase, or initial ANC <0.5 × 10^9/L increased by at least 0.5 × 10^9/L after treatment, or initial PLT <20 × 10^9/L increased by at least 20 × 10^9/L after treatment.
Overall response rate (ORR) | 6 months
  Overall response rate (ORR) was defined as the ratio of complete response (CR) + partial response (PR).CR was defined as a haemoglobin level ≥120 g/L, neutrophil count >1.5 × 10^9/L and platelet count >150 × 10^9/L in patients who did not receive a transfusion.PR was defined as not being transfusion-dependent (if previously transfusion-dependent), or doubling or normalisation of at least one cell line or baseline increase, or initial ANC <0.5 × 10^9/L increased by at least 0.5 × 10^9/L after treatment, or initial PLT <20 × 10^9/L increased by at least 20 × 10^9/L after treatment.
CRR | 3 months
  CR was defined as a haemoglobin level ≥120 g/L, neutrophil count >1.5 × 10^9/L and platelet count >150 × 10^9/L in patients who did not receive a transfusion.
CRR | 6 months
  CR was defined as a haemoglobin level ≥120 g/L, neutrophil count >1.5 × 10^9/L and platelet count >150 × 10^9/L in patients who did not receive a transfusion.

SECONDARY OUTCOMES:
safety events | 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
safety events | 6months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young NS. Aplastic anaemia. Lancet. 1995 Jul 22;346(8969):228-32. doi: 10.1016/s0140-6736(95)91273-8. No abstract available. PMID 7616805
- [Background] Young NS. Aplastic Anemia. N Engl J Med. 2018 Oct 25;379(17):1643-1656. doi: 10.1056/NEJMra1413485. No abstract available. PMID 30354958
- [Background] Bacigalupo A. How I treat acquired aplastic anemia. Blood. 2017 Mar 16;129(11):1428-1436. doi: 10.1182/blood-2016-08-693481. Epub 2017 Jan 17. PMID 28096088
- [Background] Yang C, Zhang X. Incidence survey of aplastic anemia in China. Chin Med Sci J. 1991 Dec;6(4):203-7. PMID 1813058